CLINICAL TRIAL: NCT01223196
Title: Effect of Pioglitazone on Tissue Inhibitor of Metalloproteinases 3 (TIMP-3) and TNF (Tumor Necrosis Factor)-α Converting Enzyme (TACE) in Skeletal Muscle and Their Circulating Substrates.
Brief Title: Effect of Pioglitazone on TIMP-3 and TACE in Type 2 Diabetes
Acronym: PIO-TACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Franco Folli, MD, Professor of Medicine, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HSC20080452
Record Dates: First submitted 2010-07-21; First posted 2010-10-18 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes, Thiazolidinediones, TIMP-3, TACE, TNF-a,; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): One arm of the study subjects will be treated with Placebo only, once a day, for 6 months
  Interventions: Drug: Placebo
- Pioglitazone (Active Comparator): One arm of the study subjects will be treated with Pioglitazone, 15mg, once a day, for 6 months
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — This study will examine the effect of Pioglitazone on tissue inhibitor of metalloproteinases (TIMP-3) and on TNF-alfa converting enzyme in the skeletal muscle of type 2 diabetic subjects.
  Other Names: ACTOS
  Arms: Pioglitazone
Drug: Placebo — Inactive placebo for comparison to Pioglitazone on tissue inhibitor of metalloproteinases (TIMP-3) and on TNF-alfa converting enzyme in the skeletal muscle of type 2 diabetic subjects.
  Arms: Placebo

SUMMARY:
Background: Pioglitazone has been shown to have potent anti-inflammatory as well anti-atherosclerotic effects. However, the mechanisms by which pioglitazone exerts these effects are not clear. The investigators propose that Tissue Inhibitor of MetalloProteinase-3 (TIMP-3) and TNF-alfa converting enzyme (TACE) play a major role in pioglitazone mediated improvement in insulin sensitivity and endothelial function. In animal models, low dose pioglitazone inhibits lesion progression and matrix metalloproteinase expression in advanced atherosclerotic plaques. The investigators believe that a lower dose of Pioglitazone will also have anti-inflammatory effects.

Aim: To examine the effect of low dose Pioglitazone (15mg/day) on TIMP and TACE in Pioglitazone mediated improvements in insulin sensitivity.

Methods: Thirty subjects with T2DM will participate in following studies: (i) oral glucose tolerance test (OGTT); (ii) Dual energy absorptiometry(DXA) for body fat content, (iv) skeletal muscle biopsy. Subjects will be randomized to receive either placebo or pioglitazone for 24 weeks. The investigators will study the effect of Pioglitazone on (1) TIMP and TACE substrate activity in skeletal muscle, adipose tissue, mononuclear cells, and their relationship to insulin sensitivity and vascular reactivity, other adipocytokines- resistin, TNF-α and Visfatin; (2) markers of inflammation and atherosclerosis- C-reactive protein, VCAM-1 (vascular cell adhesion molecule 1), ICAM-1 (Intercellular Adhesion Molecule 1), endothelin 1, E-selectin, P-selectin, TNFrecI (Tumor Necrosis Factor Receptor I), TNFrecII (Tumor Necrosis Factor Receptor II), IL-6 (Interleukin 6) receptor.

DETAILED DESCRIPTION:
Pioglitazone has been shown to have potent anti-inflammatory as well anti-atherosclerotic effects. However, the mechanisms by which pioglitazone exerts these effects are not clear. We propose that tissue inhibitor of metalloproteinase-3 (TIMP-3) and TNF-alfa converting enzyme (TACE) play a major role in pioglitazone mediated improvement in insulin sensitivity and endothelial function. In animal models, low dose pioglitazone inhibits lesion progression and matrix metalloproteinase expression in advanced atherosclerotic plaques. We believe that a lower dose of Pioglitazone will also have anti-inflammatory effects without the potential adverse effects of weight gain.

In order to examine the effect of low dose Pioglitazone (15mg/day) on TIMP-3 and TACE in Pioglitazone mediated improvements in insulin sensitivity and endothelial function, we propose to study subjects with type 2 diabetes mellitus (T2DM) will participate in following studies: (i) OGTT; (ii) DXA for body fat content, (iii) euglycemic hyperinsulinemic clamp, (iv) skeletal muscle biopsy.

This study will examine the effect of Pioglitazone on (1) TIMP and TACE substrate activity in skeletal muscle and their relationship to insulin sensitivity and adipocytokines- resistin, TNF-α and Visfatin; (2) markers of inflammation and atherosclerosis- C-reactive protein, VCAM-1, ICAM-1, endothelin 1, E-selectin, P-selectin, TNFrecI, TNFrecII, IL-6 rec. Fifteen subjects will receive placebo and 15 will receive pioglitazone.

Study Design.

Double blind placebo controlled parallel design.

ENDPOINTS

PRIMARY: Reduction in TIMP-3 and TACE gene expression and TACE substrate activity in skeletal muscle and adipose tissue..

SECONDARY: Improvement in: (1) Skeletal muscle insulin sensitivity, (2) plasma FFA (Free Fatty Acid) and lipid levels (3) reduction in VCAM and ICAM concentrations.

RESEARCH PLAN - EXPERIMENTAL PROTOCOL Subjects - We plan to study subjects with T2DM (BMI 30-40 Kg/m2, age=18-70 years, HbA1c <10%); of which equal number of subjects in each group will receive placebo/study drug. With this study design, we will be able to discriminate the effects of pioglitazone on TIMP3 and TACE substrate activity and gene expression in patients with T2DM and non-diabetic subjects with metabolic syndrome. Subjects in both arms of the study (placebo and study drug) will be matched for age, BMI and HbA1c and the effects of Pioglitazone in these subjects will be independent of the glucose lowering effect of the drug. Diabetic subjects who have previously received insulin or who are taking a thiazolidinedione will be excluded. Only diabetic patients who are free of other major organ disease will be studied. Only subjects whose body weight has been stable for at least three months and who do not participate in strenuous exercise will be studied.

Prior to the start of pioglitazone all subjects will participate in the following studies:

(i) Qualification visit: Physical examination, medical history, EKG tracing, complete blood cell count, SMA 24 and lipid profile will be performed. Also, fasting levels of plasma total/HDL/LDL cholesterol, triglycerides, and markers for atherosclerosis and inflammation (CRP: C-reactive protein), and hypercoagulability (plasminogen activator inhibitor -1), adiponectin, TNF-α, and HbA1c will be measured on this day.

(ii) OGTT (75 grams) to evaluate overall glucose tolerance and insulin secretion. Biopsy of the vastus lateralis muscle will be performed 30 minutes before the start of the OGTT.

(iii) Measurement of lean body mass and fat free mass with Dual Energy Xray Absorptiometry (DXA) scan.

(iv) Brachial artery reactivity with post ischemic flow mediated vasodilation and response to sublingual Nitroglycerine will be done on the same day that DXA is done.

Upon completion of the above studies, subjects will be randomly assigned to receive either placebo or pioglitazone at a dose of 15 mg day for 24 weeks. Subjects will receive dietary counseling prior to the initiation of pioglitazone therapy and be asked to consume a standard ADA, weight maintaining diet throughout the study. Patients will be seen for follow up every 2 weeks. On each follow up visit interim medical history, blood pressure, pulse, weight and fasting plasma glucose concentration will be determined. Every 4 weeks TIMP and TACE substrate activity, adiponectin, visfatin, C-reactive protein (CRP) and markers of inflammation and atherosclerosis (VCAM-1, ICAM-1, endothelin 1, E-selectin, P-selectin) will be measured. In addition, every month we will measure HbA1c, plasma lipids and liver function tests. After 24 weeks of pioglitazone treatment all subjects will have a repeat: (i) measurement of fat and lean body mass by DXA, (ii) OGTT, (iii) vastus lateralis biopsy.

The total length of the study from the start of the pioglitazone/placebo will be 26-30 weeks. The baseline studies will be performed over a period of 1 to 4 weeks. The repeat studies will be performed during the last 24-30 weeks of pioglitazone therapy.

Methods OGTT AND PERCUTANEOUS SKELETAL MUSCLE BIOPSY

All subjects will be admitted to the General Clinical Research Center (GCRC) of the South Texas Veterans Healthcare System, Audie Murphy Division, San Antonio, Texas on the day of the study between 6:45 and 8 AM. Subjects will not be allowed to eat or drink anything after 10 PM the night before, until the study is completed. At about 7:30 AM subjects will ingest 75 grams of glucose. Plasma samples for glucose, insulin and C-peptide concentrations will be drawn at -30, -15, and 0 minutes and every 15 minutes thereafter for two hours. At 30 minutes before the start of the OGTT, a muscle biopsy of the vastus lateralis muscle will be performed. After injection of xylocaine, a 5 mm incision is made 10-15 cm above the patella, and the biopsy needle is inserted into the muscle. The needle is connected to suction, and approximately 200 mg of muscle tissue is obtained. All muscle biopsies will be stored in liquid nitrogen within 15 seconds, until processing for specific assays.

We will be able to derive from the OGTT a very reliable estimate of insulin secretion as well as insulin sensitivity by calculating the "MATSUDA" index as well as the OGIS (Oral Glucose Insulin Sensitivity) index . These indexes have been shown repeatedly to correlate extremely well with the results obtained by the euglycemic clamp.

Three to seven days later, body fat content will be determined by DXA.

EUGLYCEMIC HYPERINSULINEMIC CLAMP:

On a separate day, subjects will be admitted to the General Clinical Research Center (GCRC) of the South Texas Veterans Healthcare System, Audie Murphy Division, San Antonio, Texas, between 6:45 and 8 AM for a hyper-insulinemic euglycemic (80 mU (milli-Unit)/m2•min) clamp. Continuous indirect calorimetry (Deltatrac, Sensormedics, Anaheim, CA) will be performed for 30 minutes prior to the start of the insulin clamp, and during the 150-180 minutes period of the insulin clamp to calculate rates of glucose and lipid oxidation. After obtaining the basal samples for insulin, C-peptide, a priming dose of insulin is given for first 10 minutes which is followed by constant infusion. At 5 minutes a variable rate of glucose is infused to maintain plasma glucose at ~100mg/dl for 180minutes.

Upon completion of the above studies, all subjects (diabetics, non diabetic metabolic syndrome) will be started on pioglitazone at a dose of 15 mg day and continued for 24 weeks. Subjects will receive dietary counseling prior to the initiation of pioglitazone therapy and be asked to consume a standard ADA, weight maintaining diet throughout the study. Patients will be seen for follow up every 2 weeks. On each follow up visit interim medical history, blood pressure, pulse, weight and fasting plasma glucose concentration will be determined. Every month we will measure HbA1c, plasma lipids, liver function tests, adipocytokines, and inflammatory markers as described earlier. After 4 months of pioglitazone treatment subjects will have a repeat: (i) measurement of fat and lean body mass by DXA, (ii) OGTT with vastus lateralis biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma Glucose- 126-270
* HbA1c <10%
* Hematocrit >34%
* Serum creatinine <1.8mg/dl
* AST (aspartate aminotransferase) < 2 times upper limit of normal
* ALT (Alanine aminotransferase) < 2 time upper limit of normal
* Alkaline phosphatase <2 times upper limit of normal

Exclusion Criteria:

* Type 1 DM
* Fasting plasma glucose >270 mg/dl
* Thiazolidinedione therapy
* Insulin therapy in last 3 months
* Congestive heart failure > NYHA (New York Heart Association) class II
* History of dyspnoea on exertion
* Abnormal breath sounds
* EKG changes other than non-specific ST-T changes in the ECG (Electro-CardioGram) or LVH (Left Ventricular Hypertrophy)
* H/O Claudication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Folli, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Bartter Research Unit , ALM VA Hospital, San Antonio, Texas, United States

REFERENCES:
- [Derived] Tripathy D, Daniele G, Fiorentino TV, Perez-Cadena Z, Chavez-Velasquez A, Kamath S, Fanti P, Jenkinson C, Andreozzi F, Federici M, Gastaldelli A, Defronzo RA, Folli F. Pioglitazone improves glucose metabolism and modulates skeletal muscle TIMP-3-TACE dyad in type 2 diabetes mellitus: a randomised, double-blind, placebo-controlled, mechanistic study. Diabetologia. 2013 Oct;56(10):2153-63. doi: 10.1007/s00125-013-2976-z. Epub 2013 Jun 30. PMID 23811853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 60 patients were screened and 24 met the eligibility criteria and were randomized.
Pre-assignment Details: 36 patients did not meet the eligibility criteria and were excluded.
Groups:
- Placebo: One arm of the study subjects will be treated with Placebo only, once a day.
- Pioglitazone: One arm of the study subjects will be treated with Pioglitazone, 15mg, 1 capsule/day.
Period: Overall Study
Arm/Group | Placebo | Pioglitazone
Started | 13 | 11
Completed | 9 | 11
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: One arm of the study subjects will be treated with Placebo only.
- Pioglitazone: One arm of the study subjects will be treated with Pioglitazone
- Total: Total of all reporting groups
Arm/Group | Placebo | Pioglitazone | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7) | 56.6 (9.3) | 55.7 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Whole Body Insulin Sensitivity During the Euglycemic Insulin Clamp
Description: Insulin sensitivity was measured by the euglycemic clamp before and 6 months after PIO (PIOGLITAZONE) or PLAC (PLACEBO) treatment.
  The outcome measure is Insulin sensitivity obtained from euglycemic insulin clamp and it is called M/I, where M = whole body glucose uptake during the euglycemic insulin clamp and I = circulating insulin levels during the euglycemic insulin clamp. It is expressed as Mg. of glucose/kg body weight/mU (milli Unit)x l (liter).of insulin (Ins)
Time Frame: 6 months
Population: M/I
Measure: Mean (Standard Error); unit: Mg. of glucose/kg body w./mUxl ins.
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 9 | 11
Mg. of glucose/kg body w./mUxl ins.
  M/I at baseline | 3.2 (0.01) | 3.01 (0.02)
  M/I after 6 months of treatment | 3.4 (0.02) | 3.7 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Pioglitazone; Mann-Whitney test was used to test differences in whole body insulin sensitivity (M/I) between groups. Treatment-induced changes were examined by Wilcoxon's rank test. Data were analyzed using SPSS 20 (Statistical Package for Social Sciences 20), Chicago, IL, USA); Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney); Mann-Whitney test was used to test differences in M/I. Statistical Analysis applies to (M/I) between Pioglitazone and Placebo after 6 months
Statistical Analysis 2: Comparison: Placebo vs Pioglitazone; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney); Mann-Whitney test was used to test differences in whole body insulin sensitivity (M/I) between groups

2. Secondary Outcome: Effect of Pioglitazone on TNF (Tumor Necrosis Factor) Alpha Converting Enzyme (TACE) Activity in Skeletal Muscle.
Description: The activity of TACE is measured by detecting the release of a fluorogenic synthetic substrate of TACE and measuring in a fluorometer. It is expressed in Fluorescence Units (F.U.)
Time Frame: 6 months
Population: These individuals completed both the baseline and all intermediate and the end of study visits.
Measure: Mean (Standard Error); unit: Tace Activity in F.U./mg prot
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 9 | 11
Tace Activity in F.U./mg prot
  TACE Activity at baseline (F.U./mg/prot) | 0.2 (0.03) | 0.28 (0.04)
  TACE Activity after 6 months(F.U./mg/prot) | 0.15 (0.02) | 0.06 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Pioglitazone; Mann-Whitney test was used to test differences in TACE activity in skeletal muscle between groups. Treatment-induced changes were examined by Wilcoxon's rank test. Data were analyzed using SPSS 20 (Statistical Package for Social Sciences, Chicago, IL, USA); Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mann-Whitney test was used to test differences in TACE activity in skeletal muscle between groups
Statistical Analysis 2: Comparison: Placebo vs Pioglitazone; Statistical analysis 2 also used 2-sided t-test similar to Statistical analysis -1; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Statistical Analysis applies toTNF (Tumor Necrosis Factor) alpha converting enzyme (TACE) activity between Pioglitazone and Placebo after 6 months

3. Other Pre Specified Outcome: Percentage (%) of Haemoglobin A1C
Description: HbA1c (Haemoglobin A1c) is glycosylated haemoglobin, measured as a % of total Hb in red blood cells by a standard biochemical method (HPLC).
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Percentage (%) of HbA1c
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 9 | 11
Percentage (%) of HbA1c
  HbA1c - baseline | 8.0 (0.5) | 7.0 (0.2)
  HbA1c- after 6 months | 7.7 (0.5) | 6.5 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Pioglitazone; Mann-Whitney test was used to test differences Haemoglobin A1C between groups. Treatment-induced changes were examined by Wilcoxon's rank test. Data were analyzed using SPSS 20 (Statistical Package for Social Sciences, Chicago, IL, USA); Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mann-Whitney test was used to test differences in Heamoglobin A1c between groups

ADVERSE EVENTS:
Arm/Group | Placebo | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 1/13 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Pioglitazone (N=11)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — patient was on placebo, but was noted to have marked anemia while on the study and was disenrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No